CLINICAL TRIAL: NCT02847052
Title: Study of the Role of Soluble Inhibitor of Interleukin 22, Interleukin 22 Binding Protein (IL-22BP), in Chronic Inflammatory Bowel Disease
Acronym: IL-22BP MICI
Status: Terminated | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0042
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study

SUMMARY:
IL-22 is an IL-10 family cytokine that plays major actions to increase intestinal epithelial barrier function and regeneration during experimental colitis. IL-22 binding protein is a small, soluble, and secreted protein potently inhibiting IL-22 actions through preventing the binding with IL-22 Recepteur. This study aims at characterizing how IL-22 binding protein is regulated in Inflammatory bowel disease to better understand the way IL-22 acts on epithelial cells during flares of the disease.

ELIGIBILITY:
Inclusion criteria

1. Crohn's disease or Ulcerative colitis
2. Healthy controls paired for age and sex
3. Samples availability in the biobank
4. Signed consent
5. No (Immune Mediated Inflammatory Disorders other than Inflammatory bowel disease
6. No other conditions predicted or known to affect IL-22/IL-22 recepteur /IL-22 binding protein regulation
7. Availability of clinical data
8. Age >18 y.o.
9. No pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease, Retrospective, controlled, open, monocentric study
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Regulation of Interleukine 22 binding protein expression in Crohn's disease or Ulcerative colitis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jérome Martin, Principal Investigator — Nantes University Hospital